CLINICAL TRIAL: NCT06991478
Title: A Single-arm, Prospective, Open-label, Phase I/II Study of Allogeneic NK Cell Injection (SK-NK Injection) in the Treatment of Patients With Advanced or Metastatic Malignant Solid Tumors Accompanied by Malignant Ascites
Brief Title: SK-NK Injection in Patients With Advanced Solid Tumors Accompanied by Malignant Ascites
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SK-NK-001
Record Dates: First submitted 2025-05-18; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor, Malignant Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1:Dose escalation stage (Experimental): "3+3" design. SK-NK injection, Two dose groups, namely 20×108 cells and 30×108 cells.
  Interventions: Drug: SK-NK injection
- Phase 2:Expansion stage (Experimental): The dose of SK-NK injection selected based on the results of the first stage
  Interventions: Drug: SK-NK injection

INTERVENTIONS:
Drug: SK-NK injection — In this stage, two dose groups are preset, namely 20×108 cells and 30×108 cells. Subjects who meet the inclusion criteria will receive intravenous infusion of SK-NK injection once a week for six consecutive times. After completing six consecutive infusions of SK-NK injection, the researchers evaluated that the patient benefited and could continue to receive six consecutive infusions of SK-NK injection. After completing twelve infusions, the decision on whether to continue the treatment subsequently could be made based on the patient's condition
  Arms: Phase 1:Dose escalation stage
Drug: SK-NK injection — Based on the dose selected from the results of the first stage, the clinical efficacy, safety, tolerability and pharmacokinetic characteristics of RP2D were further verified. The types of cancer and the number of cases enrolled in stage II are to be determined
  Arms: Phase 2:Expansion stage

SUMMARY:
This study is divided into two phases. Patients with recurrent or metastatic solid tumors accompanied by malignant ascites who have failed previous standard treatments are enrolled. The first phase is a single-arm, open-dose exploratory Phase I clinical study. In this phase, two dose groups are preset, namely 20×108 cells and 30×108 cells. Subjects who meet the inclusion criteria will receive intravenous infusion of SK-NK injection. Once a week for 6 consecutive infusions. After completing 6 consecutive infusions of SK-NK injection, the researchers evaluated that the patient benefited and could continue to receive 6 consecutive infusions of SK-NK injection. After completing 12 infusions, whether to continue the treatment subsequently could be determined based on the patient's condition. The second stage will be based on the results of the first stage to further verify the clinical efficacy, safety, tolerability and pharmacokinetic characteristics of RP2D, etc.

ELIGIBILITY:
Inclusion Criteria：

1. Aged 18 to 75 years.
2. Malignant solid tumors confirmed by histology or pathology, including: advanced gastric cancer, colorectal cancer, esophageal squamous cell carcinoma, gynecological malignancies, etc. that have failed at least two lines of treatment.
3. Pathological diagnosis or clinical diagnosis combined with malignant ascites, and ascites drainage is not required within one week before the administration of the study.
4. At least one measurable tumor lesion based on RECIST V1.1 criteria.
5. ECOG PS ≤1.
6. Expected survival ≥12 weeks.
7. Adequate organ function.
8. Non-reproductive female patients, or reproductive female patients whose pregnancy test results are negative and commit to taking adequate and effective contraceptive measures or abstinence from the screening period until 3 months after the last administration, or male patients commit to taking adequate and effective contraceptive measures or abstinence from the screening period until 3 months after the last administration.
9. Understands and provides written informed consent and willing to follow the requirements specified in protocol.

Exclusion Criteria:

1. History of severe allergic reactions to protein drugs
2. Have received NK cell therapy in the past.
3. Untreated, unstable or uncontrolled central nervous system (CNS) metastases.
4. Tumor invasion of vital arteries resulting in high risk of bleeding, significant risk of perforation or already formed fistulae.
5. Major surgeries within 4 weeks before enrollment or are planned to undergo major surgeries during the trial (excluding exploration surgeries).
6. New infections or concurrent infections occurred within 14 days before enrollment and have not yet been controlled to clinical stability.
7. Prior to the first study dose, systemic chemotherapy and anti-tumor monoclonal antibody drug therapy has been completed for at least 4 weeks; small molecule targeted drug therapy has been completed for at least 2 weeks or 5 half-lives of the drug (whichever is longer); intraperitoneal chemotherapy has been completed for at least 2 weeks; and treatment with proprietary Chinese medicines approved by the National Medicines and Pharmaceutical Administration (NMPA) as antitumor and having antitumor effects has been completed for at at least 2 weeks.
8. Patients with severe respiratory disease at the time of screening that results in respiratory failure or who, in the judgment of the investigator, are not suitable for enrollment.
9. Active autoimmune disease.except that the following are allowed to enter the screen: type I diabetes mellitus, hypothyroidism that can be controlled by replacement therapy only, and skin conditions (e.g., vitiligo, psoriasis, or alopecia areata) not requiring systemic therapy.
10. Patients had severe cardiovascular disease at screening, with an acute cardiovascular event or pulmonary embolism within the last 6 months or vascular stenting within 6 months; or venous thrombotic disease, such as lower extremity venous thrombosis, within the last 1 month.
11. Intestinal obstruction or gastrointestinal bleeding within 30 days prior to enrollment.
12. Objective reasons for not being able to drain ascites adequately (including segregation of ascites) or in combination with coeliac ascites.
13. Confirmed portal vein embolism or portal hypertension on examination.
14. Active chronic hepatitis B, active hepatitis C, positive human immunodeficiency virus (HIV) antibodies or active syphilis infection.
15. Combined with pleural effusion and causing clinical symptoms such as chest tightness and dyspnea, requiring clinical intervention as assessed by the investigator; or combined with moderate or greater amounts of pericardial effusion and clinical symptoms.
16. Pregnant or lactating women.
17. Subjects who, in the judgment of the investigator, have a history of other serious systemic disease or are unfit to participate in this trial for any other reason (the presence of psychiatric disorders, alcohol, drug, or substance abuse in the patient that may affect compliance with the trial, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
SK-NK injection safety and tolerance | up to 12 months
  The incidence of DLT,TEAEs and SAE, and the safety indicators before and after administration
ORR | up to 12 months
  Antitumor efficacy of SK-NK injection

SECONDARY OUTCOMES:
Pharmacokinetic (PK) characteristics of SK-NK injection; | up to 12 months
  To evaluate the Cmax of SK-NK injection in patients with advanced or metastatic malignant solid tumors accompanied by malignant ascites
DCR | up to 12 months
  Disease control rate of SK-NK injection
PFS | up to 12 months
  Progression-free survival of SK-NK injection
OS | up to 12 months
  The overall survival of the enrolled patients
Pharmacokinetic (PK) characteristics of SK-NK injection | up to 12months
  To evaluate the t1/2 of SK-NK injection in patients with advanced or metastatic malignant solid tumors accompanied by malignant ascites
Pharmacokinetic (PK) characteristics of SK-NK injection; | up to 12months
  To evaluate the Tmax of SK-NK injection in patients with advanced or metastatic malignant solid tumors accompanied by malignant ascites
Pharmacokinetic (PK) characteristics of SK-NK injection; | up to 12months
  To evaluate the AUC0-last of SK-NK injection in patients with advanced or metastatic malignant solid tumors accompanied by malignant ascites

IPD SHARING:
Plan to Share IPD: No